CLINICAL TRIAL: NCT03914573
Title: Observational Study of the Association of Participation in High School Football on Health in Late Adulthood
Brief Title: High School Football and Adult Health
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 833020
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Health Impairment; Pain; Obesity
Keywords: health; football; pain; obesity
MeSH Terms: conditions — Pain; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to determine the effect of playing high school football on self-rated health in late adulthood. This is an observational study that will use data from the Wisconsin Longitudinal Study, a longitudinal cohort of high school graduates from 1957, to compare graduates who played high school football with comparable graduates who did not play football on self-rated health, pain, functional ability, and weight at the age of 65 years.

DETAILED DESCRIPTION:
Data will be used from the Wisconsin Longitudinal Study (WLS), a long-term study of a random sample of 10,317 men and women who graduated from Wisconsin high schools in 1957 to determine the association between participation in high-school football and self-rated health, pain, and obesity in late adulthood. The WLS is an optimal observational dataset to answer these hypotheses. WLS captures early-life exposures that are important predictors of health and well-being in later life such parental socioeconomic status, occupation, and education level, family structure, and race. It also captures whether study participants participated in high school football and contains detailed measurements of their health in adulthood. WLS provides a robust and longitudinal dataset, overcoming the limitations of prior cross-sectional studies, to compare the health in later adulthood of those who played high school football to those who did not, after carefully controlling for a potential confounders

A matched observational study will be conducted, in which football players and controls will be divided into smaller subgroups which are relatively homogeneous along a range of baseline covariates. The outcomes will be compared within each matched set, after adjusting for residual imbalances in the distribution of these baseline covariates between the football players and controls.

ELIGIBILITY:
Inclusion Criteria:

• Male

Exclusion Criteria:

* No yearbook information available to determine football playing status
* Sports participation in yearbook was not recorded under senior photo or in an index
* Played a high contact sport other than football (e.g. hockey)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Graduates of Wisconsin high schools in 1957. The data comes from the Wisconsin Longitudinal Study (WLS), a long-term study of a random sample of 10,317 men and women who graduated from Wisconsin high schools in 1957.
Sampling Method: Probability Sample
Enrollment: 3355 (Actual)
Dates: Start 1957-01 (Actual); Primary Completion 2003-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Self-rated Health | Collected in 2003-2005 when participants were aged 65
  Subjects reported whether their health was excellent, very good, good, fair, or poor. We dichotomized subjects' responses, coding "excellent", "very good", and "good" as 0 and coding "fair" and "poor" as 1

SECONDARY OUTCOMES:
Pain that limits activities | Collected in 2003-2005 when participants were aged 65
  Subjects reported whether during the past 4 weeks, how many of their activities were limited by pain or discomfort. We coded subject responses as 1 if they responded that some, most, or all of their activities were limited and 0 if they responded that none or a few activities were limited.
Difficulty in Activities of Daily Living | Collected in 2003-2005 when participants were aged 65
  Subjects reported whether during the past 4 weeks, have they been able to eat, bathe, dress and use the toilet without difficulty. We coded 0 for no difficulty and 1 for any difficulty.
Maximum Lifetime Body Mass Index | Collected in the WLS mail survey in 2004
  Subjects reported their maximum lifetime weight and the age at which they weighed the most. From these responses, we computed the maximum adult BMI for each subject who reported that they reached their maximum weight when they were 18 years old or older.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gaulton, MD, Principal Investigator — University of Pennsylvania; Sameer Deshpande, PhD, Principal Investigator — Massachusetts Insitute of Technology; Dylan Small, PhD, Principal Investigator — University of Pennsylvania; Mark D Neuman, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Massachusetts Institute of Technology, Cambridge, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No